CLINICAL TRIAL: NCT00451464
Title: Studies of Apolipoprotein Genotyping on the Drug Treatment of Hyperlipidemic Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9100205283; NSC93-2314-B-002-016
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2005-07

CONDITIONS: Hyperlipidemia
Keywords: Apolipoprotein, Gene polymorphism, Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Cardiovascular-related diseases have been the majorities of the leading ten causes of death in Taiwan. Atherosclerotic cardiovascular diseases are multifactorial. Some non-modifiable risk factors (e.g. genetic trait) may attenuate the benefit of risk modification of the modifiable factors (e.g. the effect of drug treatment). Genetic epidemiology has being widely used to analyze the underline risk of cardiovascular diseases and to point the direction of treatment or prevention.

Lipoprotein is composed of lipid and protein. The genetic variation or mutation of apolipoprotein, the protein of lipoprotein, has been linked to some lipid abnormality resulting severe atherosclerotic cardiovascular diseases. ApoA-I, apo A-II, apo A-IV, apo B100, apo B48, apo C-I, apo C-II, apo C-III, apo D, and apo E are currently thought to affect lipid abnormalities. In addition, it has been documented that genetic variations are presented among different races. Apolipoprotein genetic variations or genetic polymorphism study has been emerged as an important role in the field of genetic therapy. The purpose of this 3-year study is to continue the lipid study in our laboratory, identifying the apolipoprotein genotyping in our pooled hyperlipidemic patients and normal control subjects living in Taiwan. We will observe the incidence and link apo A-I, apo A-II, apo A-IV and apo C-III genetic variations to the related lipid abnormality and cardiovascular diseases. The changes of genotyping after lipid lowering drug treatment using statin or fibrate in hypercholesterolemic or hypertriglyceridemic patients is another goal of this project.

DETAILED DESCRIPTION:
Cardiovascular-related diseases have been the majorities of the leading ten causes of death in Taiwan. Atherosclerotic cardiovascular diseases are multifactorial. Some non-modifiable risk factors (e.g. genetic trait) may attenuate the benefit of risk modification of the modifiable factors (e.g. the effect of drug treatment). Genetic epidemiology has being widely used to analyze the underline risk of cardiovascular diseases and to point the direction of treatment or prevention.

Lipoprotein is composed of lipid and protein. The genetic variation or mutation of apolipoprotein, the protein of lipoprotein, has been linked to some lipid abnormality resulting severe atherosclerotic cardiovascular diseases. ApoA-I, apo A-II, apo A-IV, apo B100, apo B48, apo C-I, apo C-II, apo C-III, apo D, and apo E are currently thought to affect lipid abnormalities. In addition, it has been documented that genetic variations are presented among different races. Apolipoprotein genetic variations or genetic polymorphism study has been emerged as an important role in the field of genetic therapy. The purpose of this 3-year study is to continue the lipid study in our laboratory, identifying the apolipoprotein genotyping in our pooled hyperlipidemic patients and normal control subjects living in Taiwan. We will observe the incidence and link apo A-I, apo A-II, apo A-IV and apo C-III genetic variations to the related lipid abnormality and cardiovascular diseases. The changes of genotyping after lipid lowering drug treatment using statin or fibrate in hypercholesterolemic or hypertriglyceridemic patients is another goal of this project.

Our results showed ApoC-III (3175NT C→G) mutation was significantly related to hypertriglyceridemia, the same relation was also found in the Apo B exon 29 (13132 NT C→G; 4311 AA Asn →Ser) mutation. It is interesting to find some hot spot mutation among Caucasian population, such as Apo B exon 26 (10699 NT C→A; 3500 AA Arg →Gln), Apo A-IV (1527-2345 NT) and Apo E exon 2 mutations, were not found in tested samples. Most of presented allele frequencies in apolipoteins genes were different between our population and Caucasian population. The present results strongly suggest that it is necessary to establish our own genetic data which are linked to diseases.

ELIGIBILITY:
Inclusion Criteria:

* Hyperlipidemia

Exclusion Criteria:

* Liver and kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2002-01; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Chen Ming-Fong, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Pan-Chyr Yang, Taipei, Taiwan